CLINICAL TRIAL: NCT03457584
Title: Effect of Air-tamponade on Intraretinal Cystoid Changes After Vitrectomy With Membrane Peeling
Brief Title: Effect of Air-tamponade on Intraretinal Cystoid Changes After Membrane Peeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cysMP
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSS arm (Active Comparator): BSS is given at the end of surgery
  Interventions: Procedure: BSS arm
- air arm (Experimental): air-tamponade is given at the end of surgery
  Interventions: Procedure: air arm

INTERVENTIONS:
Procedure: air arm — epiretinal membranes are excised during membrane peeling and air-tamponade is left in the eye
  Arms: air arm
Procedure: BSS arm — epiretinal membranes are excised during membrane Peeling and BSS is left in the eye
  Arms: BSS arm

SUMMARY:
Patients with intraretinal cystoid changes before scheduled membrane peeling for epiretinal membranes are included. Patients are randomized for balanced salt solution (BSS) or air-tamponade.

DETAILED DESCRIPTION:
Patients with intraretinal cystoid changes before scheduled membrane peeling for epiretinal membranes are included. 23G-pars plana vitrectomy with membrane peeling is performed in all patients. Before surgery patients are randomized for BSS or air-tamponade. Optical coherence tomography (OCT) is performed 5 days after and 3 months after surgery, visual acuity is measured 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* epiretinal membranes and intraretinal cystoid changes

Exclusion Criteria:

* macular edema due to other reason than epiretinal membrane
* hereditary ocular disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
resorption of intraretinal cystoid changes after surgery | 3 months
  occurrence of intraretinal cystoid changes will be diagnosed by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof, Principal Investigator — VIROS at Hanuschkrankenhaus Vienna
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria